CLINICAL TRIAL: NCT01728792
Title: Impact of Subcutaneous Versus Intramuscular Administration of Inviragen's Live Attenuated Dengue Vaccine on Safety and Immunogenicity
Brief Title: Impact of SC vs IM Administration of DENVax (TDV) on Safety and Immunogenicity
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Collaborators: Walter Reed Army Institute of Research (WRAIR) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: INV-DEN-105; U1111-1181-0251 (Registry Identifier: WHO)
Record Dates: First submitted 2012-10-16; First posted 2012-11-20 (Estimated); Results first posted 2017-01-04 (Estimated); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: Dengue Fever
Keywords: Prophylactic vaccination
MeSH Terms: conditions — Dengue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Group 1: TDV SC_2 Doses Day 0 (Experimental): Takeda's Tetravalent Dengue Vaccine Candidate (TDV), 0.5 mL, subcutaneous (SC) injection, one dose in each arm, Day 0 using a needle/syringe.
  Interventions: Biological: TDV
- Group 2: TDV IM_2 Doses Day 0 (Experimental): TDV, 0.5 mL, intramuscular (IM) injection, one dose in each arm, Day 0 using a needle/syringe.
  Interventions: Biological: TDV
- Group 3: TDV IM_2 Doses Days 0 and 90 (Experimental): TDV, 0.5 mL, IM injection, one dose on Day 0 and one dose on Day 90 using a needle/syringe.
  Interventions: Biological: TDV
- Group 4: TDV SC_2 Doses Day 0 (Experimental): TDV, 0.5 mL, SC injection, one dose in each arm, Day 0 using the PharmaJet Stratis™ device.
  Interventions: Biological: TDV
- Group 5: TDV IM_2 Doses Day 0 (Experimental): TDV, 0.5 mL, IM injection, one dose in each arm, Day 0 using the PharmaJet Stratis™ device.
  Interventions: Biological: TDV

INTERVENTIONS:
Biological: TDV — TDV IM or SC injection
  Other Names: DENVax

SUMMARY:
This study assessed the safety and immunogenicity of Takeda's Tetravalent Dengue Vaccine Candidate (TDV) previously referred to as DENVax of various dosing schedules via subcutaneous (SC) or intramuscular (IM) administration with needle/syringe or needle-free injector (PharmaJet Stratis™).

DETAILED DESCRIPTION:
The vaccine tested in this study was TDV. TDV was tested to assess safety and immunogenicity of various dosing schedules, routes of administration, and delivery methods in healthy flavivirus-seronegative adults living in a dengue non-endemic country.

The study enrolled 80 participants. Participants were randomly assigned to one of the five treatment groups:

* Group 1: TDV SC injection on Day 0 in each arm using needle/syringe
* Group 2: TDV IM injection on Day 0 in each arm using needle/syringe
* Group3: TDV IM injection on Days 0 and 90 using needle/syringe
* Group 4: TDV SC on Day 0 in each arm using the PharmaJet Stratis™ device
* Group 5: TDV IM on Day 0 in each arm using the PharmaJet Stratis™ device

This single-center trial was conducted in the United States. The overall time to participate in this study was up to 5 months. Participants made multiple visits to the clinic including a final visit at Day 120 for a safety follow-up assessment.

This work was supported by the US Army Medical Research and Materiel Command under Contract No. W81XWH-12-C-0278.

The views, opinions and/or findings contained in this report are those of the author(s) and should not be construed as an official Department of the Army position, policy or decision unless so designated by other documentation.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women at least 18 years and ≤ 45 years of age at time of screening.
2. In good health as determined by medical history and physical examination (including blood pressure and heart rate).
3. Weight: Body Mass Index (BMI) ≤ 35.
4. Blood tests negative for antibodies to human immunodeficiency virus-1 (HIV-1), Hepatitis C, and Hepatitis B surface antigen.
5. Females who are not surgically sterile or post-menopausal must have a negative urine pregnancy test immediately prior to vaccination and be willing to use oral, implantable, transdermal or injectable contraceptives or another reliable means of contraception approved by the Investigator (intrauterine device, female condom, diaphragm with spermicidal foam, cervical cap, use of condom by the sexual partner or a sterile sexual partner, or abstinence) from screening until the blood sample on Day 120.
6. Willing and able to give written informed consent to participate.
7. Willing and able to communicate with the Investigator and understand the requirements of the study.
8. Access to a fixed or mobile telephone.

Exclusion Criteria

1. Any condition which would limit the participant's ability to complete the study in the opinion of the Investigator.
2. Any Grade 2 or above abnormality in the screening laboratory tests.
3. Febrile illness (temperature ≥ 38°C or 100.4°F) or moderate or severe acute illness or infection within three days before vaccination.
4. History of any significant dermatologic disease in the last 6 months, particularly with a maculopapular or petechial rash. However, if a participant had a self-limited Candida infection that was cured, then the participant can be enrolled if there is no evidence of an infection for at least 3 weeks prior to the date of dosing. If the participant has acne limited to the face, topical medications are allowed except for 2 weeks prior and 4 weeks after each dose. Oral medications for acne are excluded for 1 month prior to the start of dosing.
5. History of dengue fever, Japanese encephalitis, West Nile, or Yellow Fever disease.
6. Seropositivity to dengue or West Nile (WN) virus.
7. History of travel to dengue endemic areas including the Caribbean, Mexico, Central America, South America or Southeast Asia during the month prior to screening, or planned travel to a dengue endemic area during the study period.
8. Extensive scarring or tattoo (> 50%) on arms, shoulders, neck, face and head that could identify a participant in photos or hinder the evaluation of injection site reactions. In addition, no tattoo on the arms is permitted during the study and for one month after the final injection.
9. History of recurring headaches or migraines (more frequent than once per week) or on prescription medication for treatment of recurring headaches or migraines.
10. Hypersensitivity to any vaccine.
11. Receipt or planned receipt of any vaccine in the 4 weeks preceding or following the Day 0 or 90 injections.
12. Previous vaccination (in a clinical trial or with an approved product) against yellow fever (YF) or Japanese Encephalitis (JE).
13. Known or suspected congenital or acquired immunodeficiency or immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within the preceding 6 months.
14. Use of systemic corticosteroids therapy within the previous 6 months (at a dose of at least 0.5 mg/kg/day prednisone equivalent). Topical prednisone is not permitted if currently in use or used within the last month. Inhaled prednisone is permitted.
15. Use of any non-steroidal anti-inflammatory drugs (NSAIDs), acetaminophen or antihistamines for the 3 days immediately prior to each vaccination.
16. History of diabetes mellitus.
17. History of thymic pathology, thymectomy, myasthenia or any immunodeficiency.
18. Positive urine screen for cocaine, amphetamines, opiates, or cannabinoids
19. Known history of alcohol abuse.
20. Receipt of any other investigational product or participation in any other clinical trial of a product or device within 30 days before the first vaccination (Day 0) or planned participation in any other clinical trial while enrolled in this trial (though Day 120).
21. Receipt of blood products or immunoglobulins 8 weeks before the first vaccination (Day 0) or planned use during the period of this study (through Day 120).
22. Planned donation of blood during the period of this study (through Day 120).
23. Females who are pregnant or lactating.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2013-01-22 (Actual); Primary Completion 2013-11-01 (Actual); Study Completion 2013-11-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda
Locations (1):
- SUNY Upstate Medical University, Syracuse, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 1 investigative site in the United States from 22 January 2013 to 21 November 2013.
Pre-assignment Details: Healthy participants were randomized equally to 1 of 5 TDV treatment groups: 2 doses subcutaneous (SC) on Day 0 using needle/syringe, 2 doses intramuscular (IM) on Day 0 using needle/syringe, 1 dose IM on Days 0 and 90 using needle/syringe, 2 doses SC on Day 0 using the PharmaJet Stratis™ device and 2 doses IM on Day 0 using the PharmaJet Stratis™.
Groups:
- Group 1: TDV SC_ 2 Doses Day 0: Takeda's Tetravalent Dengue Vaccine Candidate (TDV), 0.5 mL, subcutaneous (SC) injection, one dose in each arm, Day 0 using needle/syringe.
- Group 2: TDV IM_2 Doses Day 0: TDV, 0.5 mL, intramuscular (IM) injection, one dose in each arm, Day 0 using needle/syringe.
- Group 3: TDV IM_2 Doses Days 0 and 90: TDV, 0.5 mL, IM injection, one dose on Day 0 and one dose on Day 90 using needle/syringe.
- Group 4: TDV SC_2 Doses Day 0: TDV, 0.5 mL, SC injection, one dose in each arm, Day 0 using PharmaJet Stratis™ device.
- Group 5: TDV IM_2 Doses Day 0: TDV, 0.5 mL, IM injection, one dose in each arm, Day 0 using PharmaJet Stratis™ device.
Period: Overall Study
Arm/Group | Group 1: TDV SC_ 2 Doses Day 0 | Group 2: TDV IM_2 Doses Day 0 | Group 3: TDV IM_2 Doses Days 0 and 90 | Group 4: TDV SC_2 Doses Day 0 | Group 5: TDV IM_2 Doses Day 0
Started | 14 | 16 | 17 | 17 | 16
Completed | 11 | 14 | 13 | 14 | 16
Not Completed | 3 | 2 | 4 | 3 | 0
Not completed — Withdrawal of Consent | 1 | 1 | 0 | 1 | 0
Not completed — Lost to Follow-up | 2 | 1 | 4 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set included all enrolled participants who received at least 1 dose of study vaccine and for whom any post-vaccination safety data has been obtained.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: TDV SC_ 2 Doses Day 0 | Group 2: TDV IM_2 Doses Day 0 | Group 3: TDV IM_2 Doses Days 0 and 90 | Group 4: TDV SC_2 Doses Day 0 | Group 5: TDV IM_2 Doses Day 0 | Total
Number analyzed (Participants) | 14 | 16 | 17 | 17 | 16 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.2 (5.81) | 30.2 (7.49) | 27.5 (7.92) | 30.4 (7.48) | 30.8 (7.79) | 29.4 (7.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 7 | 6 | 6 | 30
  Male | 9 | 10 | 10 | 11 | 10 | 50
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic | 0 | 1 | 2 | 1 | 0 | 4
  Non-Hispanic | 14 | 15 | 15 | 16 | 16 | 76
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 2 | 3
  Asian | 1 | 0 | 1 | 0 | 0 | 2
  Black or African American | 1 | 2 | 2 | 4 | 1 | 10
  Native Hawaiian or Pacific Islander | 1 | 0 | 0 | 0 | 0 | 1
  White | 11 | 14 | 12 | 13 | 13 | 63
  Missing | 0 | 0 | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 14 | 16 | 17 | 17 | 16 | 80

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Solicited Local (Injection Site) Reactions Following Either Vaccine Administration (Day 0 or Day 90) by Maximum Severity as Assessed by the Investigator
Description: Injection site reactions were evaluated by the investigator within 14 days following each injection. Erythema (redness), edema (swelling/induration) and pain were graded per The FDA Guidance for Industry: Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials. Pain was graded from 0=None to 4=Life-threatening. Erythema and Edema longest diameter were graded using the scale: 0=<2.5 centimeters (cm) to 3=Severe: >10 cm. Itching was graded using Common Terminology Criteria for Adverse Events (CTCAE) 4.03 where: Grade 0=no itching to Grade 3=severe. Injection site reactions are presented as the number of participants experiencing a reaction, by reaction type, overall and by severity, using the participant's worst reported severity grade. Only categories for which there was at least 1 participant are reported. Group 3 participants received 2 doses 90 days apart; injection site reactions following either vaccination are combined.
Time Frame: For 14 days after each vaccination (Up to Day 14 and/or Day 104)
Population: Safety Analysis Set included all enrolled participants who received at least 1 dose of study vaccine and for whom post-dosing data was obtained.
Measure: Number; unit: participants
Arm/Group | Group 1: TDV SC_ 2 Doses Day 0 | Group 2: TDV IM_2 Doses Day 0 | Group 3: TDV IM_2 Doses Days 0 and 90 | Group 4: TDV SC_2 Doses Day 0 | Group 5: TDV IM_2 Doses Day 0
Number analyzed (Participants) | 14 | 16 | 17 | 17 | 16
participants
  Erythema_Any Grade | 2 | 0 | 0 | 4 | 3
  Erythema_Grade 1 | 1 | 0 | 0 | 3 | 3
  Erythema_Grade 2 | 1 | 0 | 0 | 1 | 0
  Edema_Any Grade | 0 | 0 | 0 | 0 | 0
  Pain_Any Grade | 1 | 5 | 7 | 6 | 7
  Pain_Grade 1 | 1 | 5 | 6 | 5 | 7
  Pain_Grade 2 | 0 | 0 | 1 | 1 | 0
  Itching_Any Grade | 1 | 0 | 0 | 2 | 2
  Itching_Grade 1 | 1 | 0 | 0 | 0 | 1
  Itching_Grade 2 | 0 | 0 | 0 | 2 | 1

2. Primary Outcome: Number of Participants With Solicited Participant-Reported Local (Injection Site) Reactions Following Either Vaccine by Maximum Severity
Description: Injection site reactions were recorded by the participant in a memory aid for 14 days following each injection. Participants measured and recorded the longest diameter of redness (erythema) or swelling (edema) using the scale: 0=< 2.5 cm to 3= Severe: > 10 cm. For pain and itching they recorded intensity grade: 0=not present, 1=mild, 2=moderate or 3=severe. Participant-recorded local reactions are presented as number of participants reporting a reaction, by reaction type, overall and by severity, using the participant's worst reported severity grade. Only those score categories for which there was at least 1 participant are reported. Group 3 participants received 2 doses 90 days apart; injection site reactions following either vaccination are combined.
Time Frame: For 14 days after each vaccination (Up to Day 14 and/or Day 104)
Population: Participants from the Safety Analysis Set, all enrolled participants who received at least 1 dose of study vaccine and for whom post-dosing data was obtained.
Measure: Number; unit: participants
Arm/Group | Group 1: TDV SC_ 2 Doses Day 0 | Group 2: TDV IM_2 Doses Day 0 | Group 3: TDV IM_2 Doses Days 0 and 90 | Group 4: TDV SC_2 Doses Day 0 | Group 5: TDV IM_2 Doses Day 0
Number analyzed (Participants) | 14 | 16 | 17 | 17 | 16
participants
  Erythema_Any Grade (n=9,10,14,14,13) | 3 | 0 | 0 | 4 | 3
  Erythema_Grade 1 (n=9,10,14,14,13) | 2 | 0 | 0 | 2 | 2
  Erythema_Grade 2 (n=9,10,14,14,13) | 1 | 0 | 0 | 1 | 1
  Erythema_Grade 3 (n=9,10,14,14,13) | 0 | 0 | 0 | 1 | 0
  Edema_Any Grade (n=8,10,14,12,12) | 2 | 0 | 0 | 2 | 2
  Edema_Grade 1 (n=8,10,14,12,12) | 2 | 0 | 0 | 1 | 2
  Edema_Grade 2 (n=8,10,14,12,12) | 0 | 0 | 0 | 1 | 0
  Pain_Any Grade (n=13,16,17,17,16) | 10 | 7 | 8 | 11 | 10
  Pain_Grade 1 (n=13,16,17,17,16) | 7 | 7 | 8 | 9 | 7
  Pain_Grade 2 (n=13,16,17,17,16) | 3 | 0 | 0 | 2 | 3
  Itching_Any Grade (n=13,15,17,17,16) | 0 | 0 | 0 | 3 | 2
  Itching_Grade 1 (n=13,15,17,17,16) | 0 | 0 | 0 | 2 | 2
  Itching_Grade 2 (n=13,15,17,17,16) | 0 | 0 | 0 | 1 | 0

3. Primary Outcome: Number of Participants With Solicited Participant-Reported Systemic Adverse Events (AEs) Following Either Vaccine by Maximum Severity
Description: Solicited systemic AEs were recorded by the participant into a memory aid for 14 days following each vaccination. Solicited systemic AEs included: headache, muscle pain (myalgia), joint pain (arthralgia), eye pain, sensitivity to light (photophobia), tiredness (fatigue), body rash, nausea and vomiting. Systemic AEs were graded per The FDA Guidance for Industry: Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trial where: Grade 0=none to Grade 4=severe. A systemic AE of fever (defined as ≥ 100.4°F) was derived from a daily temperature reading recorded in the memory aid. Solicited systemic AEs are presented as the number of participants reporting the event, by, AE, overall and by severity, using the participant's worst reported severity grade. Group 3 participants received 2 doses 90 days apart; systemic AEs following either vaccination are combined.
Time Frame: For 14 days after each vaccination (Up to Day 14 and/or Day 104)
Population: Participants from the Safety Analysis Set included all enrolled participants who received at least 1 dose of study vaccine and for whom post-dosing data was obtained.
Measure: Number; unit: participants
Arm/Group | Group 1: TDV SC_ 2 Doses Day 0 | Group 2: TDV IM_2 Doses Day 0 | Group 3: TDV IM_2 Doses Days 0 and 90 | Group 4: TDV SC_2 Doses Day 0 | Group 5: TDV IM_2 Doses Day 0
Number analyzed (Participants) | 14 | 16 | 17 | 17 | 16
participants
  Fever_Any Grade (n=13,16,17,17,16) | 0 | 0 | 0 | 0 | 0
  Headache_Any Grade | 3 | 3 | 9 | 6 | 5
  Headache_Grade 1 | 3 | 2 | 3 | 5 | 3
  Headache_Grade 2 | 0 | 0 | 5 | 0 | 2
  Headache_Grade 3 | 0 | 1 | 1 | 1 | 0
  Myalgia_Any Grade | 2 | 2 | 3 | 3 | 2
  Myalgia_Grade 1 | 2 | 2 | 1 | 3 | 2
  Myalgia_Grade 2 | 0 | 0 | 2 | 0 | 0
  Arthralgia_Any Grade | 2 | 0 | 1 | 1 | 3
  Arthralgia_Grade 1 | 2 | 0 | 0 | 1 | 3
  Arthralgia_Grade 2 | 0 | 0 | 1 | 0 | 0
  Eye Pain_Any Grade | 0 | 0 | 0 | 0 | 0
  Photophobia_Any Grade | 2 | 1 | 4 | 0 | 2
  Photophobia_Grade 1 | 2 | 0 | 3 | 0 | 1
  Photophobia_Grade 2 | 0 | 1 | 1 | 0 | 1
  Fatigue_Any Grade | 6 | 5 | 6 | 6 | 2
  Fatigue_Grade 1 | 3 | 4 | 1 | 6 | 1
  Fatigue_Grade 2 | 3 | 1 | 5 | 0 | 0
  Fatigue_Grade 3 | 0 | 0 | 0 | 0 | 1
  Rash_Any Grade | 1 | 0 | 3 | 3 | 1
  Rash_Grade 1 | 1 | 0 | 3 | 2 | 0
  Rash_Grade 2 | 0 | 0 | 0 | 1 | 1
  Nausea_Any Grade | 3 | 3 | 4 | 2 | 3
  Nausea_Grade1 | 2 | 2 | 2 | 1 | 3
  Nausea_Grade 2 | 1 | 1 | 2 | 0 | 0
  Nausea_Grade 3 | 0 | 0 | 0 | 1 | 0
  Vomiting_Any Grade | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Participants With at Least 1 Unsolicited Related Adverse Event Following Either Vaccine Dose
Description: An Adverse Event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. The investigator assessed whether the AE was related to the study vaccination.
Time Frame: For 30 days after each vaccination for non-serious AEs and through the end of the study for SAEs (Up to 120 Days)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Group 1: TDV SC_ 2 Doses Day 0 | Group 2: TDV IM_2 Doses Day 0 | Group 3: TDV IM_2 Doses Days 0 and 90 | Group 4: TDV SC_2 Doses Day 0 | Group 5: TDV IM_2 Doses Day 0
Number analyzed (Participants) | 14 | 16 | 17 | 17 | 16
participants | 1 | 2 | 2 | 3 | 3

5. Primary Outcome: Number of Participants With at Least 1 Serious Adverse Event During the Study
Description: An Adverse Event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment.
  A serious adverse event is any experience that suggests a significant hazard, contraindication, side effect or precaution that: results in death, is life-threatening, required in-patient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect or is medically significant.
Time Frame: First Vaccination to End of Study (Up to Day 120)
Population: Safety Analysis Set includes all enrolled participants who received at least 1 dose of study vaccine and for whom post-dosing data was obtained.
Measure: Number; unit: participants
Arm/Group | Group 1: TDV SC_ 2 Doses Day 0 | Group 2: TDV IM_2 Doses Day 0 | Group 3: TDV IM_2 Doses Days 0 and 90 | Group 4: TDV SC_2 Doses Day 0 | Group 5: TDV IM_2 Doses Day 0
Number analyzed (Participants) | 14 | 16 | 17 | 17 | 16
participants | 0 | 0 | 0 | 0 | 1

6. Primary Outcome: Seroconversion Rate to Each of Four Dengue Serotypes
Description: Seroconversion rate was defined as the percentage of participants with Plaque Reduction Neutralization Test titer resulting in 50 % reduction in Plaques (PRNT50) titer ≥ 10 for participants seronegative at Baseline or a greater than four-fold increase in PRNT50 for participants seropositive at Baseline.
Time Frame: Approximately 28 to 30 days after each vaccination (Up to Day 30 and/or Day 104)
Population: Protocol deviations results in testing not performed for outcome measure.
Arm/Group | Group 1: TDV SC_ 2 Doses Day 0 | Group 2: TDV IM_2 Doses Day 0 | Group 3: TDV IM_2 Doses Days 0 and 90 | Group 4: TDV SC_2 Doses Day 0 | Group 5: TDV IM_2 Doses Day 0
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

7. Secondary Outcome: Number of Participants With Detected Viral RNA for Each TDV Component After First and Second Vaccinations
Description: Viral RNA was assessed for the four dengue components: Dengue-1 (TDV-1), Dengue-2 (TDV-2), Dengue-3 (TDV-3) and Dengue-4 (TDV-4). Only those time-points where at least 1 participant had Viral RNA detected are reported. Baseline (Day 0) and Day 7 are added for reference. "n" in each of the categories is the number of participants with data available.
Time Frame: Days 0, 7, 9, 11, 14, 17, 21, 90, 97 and 104
Population: Participants from the Safety Analysis Set, all enrolled participants who received at least 1 dose of study vaccine, with data available at the given time-point.
Measure: Number; unit: participants
Arm/Group | Group 1: TDV SC_ 2 Doses Day 0 | Group 2: TDV IM_2 Doses Day 0 | Group 3: TDV IM_2 Doses Days 0 and 90 | Group 4: TDV SC_2 Doses Day 0 | Group 5: TDV IM_2 Doses Day 0
Number analyzed (Participants) | 14 | 16 | 17 | 17 | 16
participants
  Day 0_TDV-1, TDV-2, TDV-3, TDV-4 | 0 | 0 | 0 | 0 | 0
  Day 7_TDV-1, TDV-2, TDV-3, TDV-4 (n=7,8,9,8,7) | 0 | 0 | 0 | 0 | 0
  Day 9_TDV-1, TDV-3, TDV-4 (n=6,8,7,9,9) | 0 | 0 | 0 | 0 | 0
  Day 9 _TDV-2 (n=6,8,7,9,9) | 3 | 2 | 1 | 5 | 3
  Day 11_TDV-1, TDV-3 (n=7,8,9,7,7) | 0 | 0 | 0 | 0 | 0
  Day 11_TDV-2 (n=7,8,9,7,7) | 3 | 5 | 4 | 3 | 3
  Day 11_TDV-4 (n=7,8,9,7,7) | 0 | 0 | 1 | 0 | 0
  Day 14_TDV-1, TDV-3, TDV-4 (n=6,8,7,10,9) | 0 | 0 | 0 | 0 | 0
  Day 14_TDV-2 (n=6,8,7,10,9) | 2 | 3 | 1 | 9 | 3
  Day 17_TDV-1, TDV-3, TDV-4 (n=7,8,9,8,7) | 0 | 0 | 0 | 0 | 0
  Day 17_TDV-2 (n=7,8,9,8,7) | 4 | 2 | 2 | 3 | 2
  Day 21_TDV-1, TDV-3, TDV-4 (n=6,8,8,9,9) | 0 | 0 | 0 | 0 | 0
  Day 21_TDV-2 (n=6,8,8,9,9) | 1 | 0 | 0 | 0 | 2

8. Secondary Outcome: Geometric Mean Neutralizing Antibody Titers (GMTs) of All Four Dengue Serotypes
Time Frame: Days 28, 90 and 120 after 1st vaccination
Population: Protocol deviations results in testing not performed for outcome measure.
Arm/Group | Group 1: TDV SC_ 2 Doses Day 0 | Group 2: TDV IM_2 Doses Day 0 | Group 3: TDV IM_2 Doses Days 0 and 90 | Group 4: TDV SC_2 Doses Day 0 | Group 5: TDV IM_2 Doses Day 0
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Unsolicited AEs: up to 30 days after each vaccination; SAEs: throughout the study (Up to Day 120)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study vaccine.
Arm/Group | Group 1: TDV SC_ 2 Doses Day 0 | Group 2: TDV IM_2 Doses Day 0 | Group 3: TDV IM_2 Doses Days 0 and 90 | Group 4: TDV SC_2 Doses Day 0 | Group 5: TDV IM_2 Doses Day 0
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/16 | 0/17 | 0/17 | 1/16
Other Adverse Events (participants affected / at risk) | 9/14 | 7/16 | 10/17 | 7/17 | 11/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: TDV SC_ 2 Doses Day 0 (N=14) | Group 2: TDV IM_2 Doses Day 0 (N=16) | Group 3: TDV IM_2 Doses Days 0 and 90 (N=17) | Group 4: TDV SC_2 Doses Day 0 (N=17) | Group 5: TDV IM_2 Doses Day 0 (N=16)
Cyanosis (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: TDV SC_ 2 Doses Day 0 (N=14) | Group 2: TDV IM_2 Doses Day 0 (N=16) | Group 3: TDV IM_2 Doses Days 0 and 90 (N=17) | Group 4: TDV SC_2 Doses Day 0 (N=17) | Group 5: TDV IM_2 Doses Day 0 (N=16)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Endocrine disorder (Endocrine disorders) | 0 | 1 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 1 | 0 | 0 | 0
Conjunctivitis (Eye disorders) | 0 | 0 | 0 | 1 | 0
Eye pain (Eye disorders) | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 2 | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 1 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 1 | 0 | 0
Chills (General disorders) | 0 | 0 | 1 | 0 | 0
Injection site scar (General disorders) | 0 | 0 | 0 | 1 | 0
Pain (General disorders) | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 0 | 0
Multiple allergies (Immune system disorders) | 0 | 0 | 1 | 1 | 0
Eye infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Pharyngitis streptococcal (Infections and infestations) | 0 | 1 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Tooth infection (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 2 | 2 | 2
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Vaginitis bacterial (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Viral infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Corneal abrasion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Epicondylitis (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 0 | 1 | 1 | 2
Migraine (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Glycosuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 0 | 1 | 0 | 1
Erectile dysfunction (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 1 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Ingrown hair (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
Due to protocol non-compliance issues, sponsor decided to only report safety data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No publication related to study results will be made without Sponsor's prior written approval. Any proposed publication or presentation will be submitted to Sponsor for review 60 days in advance of publication. Institution will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for an additional 60 days to preserve intellectual property.